CLINICAL TRIAL: NCT04541589
Title: A TWINSS Extension Trial to Evaluate the Safety and Tolerability of CFZ533 (Iscalimab) at Two Dose Levels Administered Subcutaneously in Patients With Sjögren's Syndrome
Brief Title: Study of Safety and Tolerability of CFZ533 in Patients With Sjögren's Syndrome
Acronym: TWINSS Extn
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCFZ533B2201E1; 2020-001942-20 (EudraCT Number)
Record Dates: First submitted 2020-08-14; First posted 2020-09-09 (Actual); Results first posted 2025-06-29 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Sjogren's Syndrome
Keywords: Sjogren's Syndrome; autoimmune; ESSDAI; ESSPRI; anti-CD40; CFZ533; iscalimab; TWINSS Extension
MeSH Terms: conditions — Sjogren's Syndrome | interventions — iscalimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study was conducted as a double-blind treatment until the final database lock of the Core study (NCT03905525). During this period, participants, Investigator, site staff, and persons performing the assessments remained blinded to the identity of the treatment until the final database lock of Core study (NCT03905525)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Iscalimab 600 mg (Experimental): Participants received 600 mg (2 injections of 300 mg/2 mL) of iscalimab subcutaneously weekly for the initial 3 weeks as loading doses, followed by a bi-weekly maintenance regimen at 600 mg (2 injections of 300 mg/2 mL).
  Interventions: Drug: Iscalimab
- Arm 2 - Iscalimab 300 mg (Experimental): Participants received one dose of 600 mg (2 injections of 300 mg/2 mL) of iscalimab subcutaneously on the first day of the extension study; then 300 mg weekly (1 injection of 300 mg/2 mL of iscalimab and 1 injection of 2 mL of placebo) for the next 2 weeks as loading doses. This was followed by a bi-weekly maintenance regimen of 300 mg (1 injection of 300 mg/2 mL of iscalimab and 1 injection of 2 mL of placebo). After the final database lock of the core study, participants underwent unblinding, leading to the discontinuation of placebo injections.
  Interventions: Drug: Iscalimab; Other: Placebo

INTERVENTIONS:
Drug: Iscalimab — Iscalimab 600 mg or 300 mg was administered subcutaneously weekly for the first 3 weeks. Subsequently, iscalimab was administered subcutaneously bi-weekly (every other week or Q2W).
  Other Names: CFZ533
Other: Placebo — Placebo (1 injection of 2 ml) administered to participants in the iscalimab 300 mg arm to maintain blinding until the final database lock of the core study
  Arms: Arm 2 - Iscalimab 300 mg

SUMMARY:
This study will evaluate the safety and tolerability of iscalimab at two dose levels in patients with Sjögren's Syndrome, who participated in the TWINSS core study, CCFZ533B2201 (NCT03905525). Additionally, this Extension study will further explore the pharmacokinetics (PK) and efficacy of iscalimab at two dose level.

DETAILED DESCRIPTION:
This study was a continuation of the TWINSS core study CCFZ533B2201 (NCT03905525) that offered continuation of treatment for participants who completed the core study and were deemed by the Investigator to clinically benefit from continued iscalimab therapy based upon response to therapy at the end of the treatment period of the core study. The extension study was a 48-week treatment study, with a safety follow-up period of 12 weeks, to provide additional safety and tolerability information for iscalimab.At Week 60 of the TWINSS core study, eligible participants had the option to enroll in the extension study.

Participants were classified as treatment responders or non-responder based on their European League Against Rheumatism (EULAR) Sjögren's syndrome disease activity index (ESSDAI) and EULAR Sjögren's syndrome patient reported index (ESSPRI) scores from predefined time points in the core study. In the extension study, participants were reassigned to either iscalimab 600 mg or 300 mg subcutaneously via prefilled syringes (PFS) based on their responder status and the iscalimab doses that they received in the core study

All participants enrolled in the extension study received a weekly loading regimen at the start of the treatment period for the initial 3 weeks, followed by a subcutaneous maintenance regimen (600 or 300 mg subcutaneously every 2 weeks). Injections were performed at site or at home by site staff or participant/caregiver.

Study blinding for the extension study was maintained until final database lock of the core study, upon which the participants and Investigators were unblinded, making it an open-label study through Week 120 (end of study visit).

ELIGIBILITY:
Inclusion Criteria:

1. Participants had to have participated in the TWINSS core study, CCFZ533B2201 (NCT03905525), and had to have completed the entire treatment period up to Week 48 and the follow-up period up to Week 60.
2. Signed informed consent had to be obtained prior to participation in the Extension study (i.e., before commencement of the Week 60 assessments of the core study).
3. In the judgment of the Investigator, participants had to be expected to clinically benefit from continued iscalimab therapy.

Exclusion Criteria:

1. Sjögren's Syndrome overlap syndromes where another autoimmune rheumatic disease constituted the principle illness, specifically:

   * Moderate-to-severe active systemic lupus erythematosus (SLE) with anti-dsDNA positivity and renal involvement, or other organ involvement that impeded on the ability to score ESSDAI domains
   * Active rheumatoid arthritis (RA) that impeded on the ability to score the ESSDAI articular domain
   * Systemic sclerosis
   * Any other concurrent connective tissue disease (e.g., lupus nephritis (LN), large vessel vasculitis (LVV), Sharp syndrome (mixed connective tissue disease) that was active and required immunosuppressive treatment outside the scope of this trial and would impede on Sjögren's Syndrome organ domain assessments
2. Use of other investigational drugs other than iscalimab during the core study
3. Active uncontrolled viral, bacterial or other infections requiring systemic treatment at the time of enrollment, or history of recurrent clinically significant infection or of bacterial infections with encapsulated organisms
4. Pregnant or nursing (lactating) women, where pregnancy was defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human Chorionic Gonadotropin (hCG) laboratory test
5. Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, unless they were using highly effective methods of contraception during dosing and for 14 weeks after stopping the investigational drug.
6. Missing ESSDAI (Cohort 1 and Cohort 2) or ESSPRI (Cohort 2) scores in the core study at Weeks 0 and 4 or Weeks 40 and 48.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (60):
- United States (7):
  - North GA Rheumatology Group PC, Suwanee, Georgia
  - Ochsner Health System, Baton Rouge, Louisiana
  - The John Hopkins Jerome L Greene Sjogren, Baltimore, Maryland
  - Tufts School of Dental Medicine, Boston, Massachusetts
  - Winthrop University Hospital, Mineola, New York
  - Perelman School of Medicine, Philadelphia, Pennsylvania
  - Uni Wisconsin School Med Pub Health, Madison, Wisconsin
- Argentina (2):
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, CABA
- Novartis Investigative Site, Nedlands, Western Australia, Australia
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Vienna
- Brazil (3):
  - Novartis Investigative Site, Vitória, Espírito Santo
  - Novartis Investigative Site, Juiz de Fora, Minas Gerais
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (3):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Rimouski, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Chile (3):
  - Novartis Investigative Site, Valdivia, Los Ríos Region
  - Novartis Investigative Site, Santiago, RM
  - Novartis Investigative Site, Santiago
- Colombia (2):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Barranquilla, Atlántico
- France (4):
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Strasbourg
- Germany (4):
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Athens, Greece
- Hungary (2):
  - Novartis Investigative Site, Székesfehérvár, Fejér
  - Novartis Investigative Site, Szeged
- Israel (3):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Ramat Gan
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pisa, PI
- Japan (4):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Sasebo, Nagasaki
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Chuo Ku, Tokyo
- Netherlands (2):
  - Novartis Investigative Site, Rotterdam, South Holland
  - Novartis Investigative Site, Groningen
- Portugal (2):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Ponte de Lima
- Romania (2):
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Cluj-Napoca
- Russia (5):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Tomsk
  - Novartis Investigative Site, Yekaterinburg
- Novartis Investigative Site, Seoul, Seocho Gu, South Korea
- Novartis Investigative Site, Stockholm, SE, Sweden
- Novartis Investigative Site, Ankara, Turkey (Türkiye)
- United Kingdom (3):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Doncaster
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: Core study — https://clinicaltrials.gov/ct2/show/NCT03905525?term=CCFZ533B2201&draw=2&rank=1
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2657

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed the core study (CCFZ533B2201, NCT03905525) and were deemed by the Investigator to clinically benefit from continued iscalimab therapy based upon response to therapy at the end of the treatment period of the core study were enrolled in this study
Period: Treatment Period
Arm/Group | Arm 1: Iscalimab 600 mg | Arm 2 - Iscalimab 300 mg
Started | 152 | 54
Completed | 133 | 47
Not Completed | 19 | 7
Not completed — Adverse Event | 8 | 2
Not completed — Physician Decision | 3 | 1
Not completed — Subject decision | 7 | 4
Not completed — Withdrawal by Subject | 1 | 0
Period: Safety Follow-up Period
Arm/Group | Arm 1: Iscalimab 600 mg | Arm 2 - Iscalimab 300 mg
Started | 152 | 54
Completed | 143 | 49
Not Completed | 9 | 5
Not completed — Adverse Event | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Subject decision | 5 | 3
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Iscalimab 600 mg | Arm 2 - Iscalimab 300 mg | Total
Number analyzed (Participants) | 152 | 54 | 206
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 126 | 45 | 171
  >=65 years | 26 | 9 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 53 | 201
  Male | 4 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 125 | 45 | 170
  Black or African American | 5 | 2 | 7
  Asian | 16 | 6 | 22
  American Indian or Alaska Native | 4 | 1 | 5
  Unknown | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence (e.g., any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a participant. TEAE included all AEs up to the last dose date plus 14 weeks or the end of the entire study (including the safety follow-up period), whichever occurred earlier. A patient with multiple severity ratings for an AE was only counted under the maximum rating. Additionally, a patient with multiple occurrences of an event was counted only once. The severity of AEs was assessed using the Common Terminology Criteria for Adverse Events, with the following grading system: Mild: usually transient in nature and generally not interfering with normal activities; Moderate: sufficiently discomforting to interfere with normal activities; Severe: prevented normal activities.
  A serious adverse event (SAE) was defined as any AE that required medical intervention, hospitalization, or results in death, disability, or a birth defect.
Time Frame: From start of extension study up to 14 weeks after last study-drug administration or end of study (whichever occurred earlier), assessed up to approximately 60 weeks
Population: The Safety Set (SAF) included all participants who received at least one dose of study treatment. Participants were analyzed according to the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Iscalimab 600 mg | Arm 2 - Iscalimab 300 mg
Number analyzed (Participants) | 152 | 54
Participants
  Death | 0 | 0
  Adverse event (all severities) | 127 | 43
  Adverse Event- Mild | 57 | 24
  Adverse Event- Moderate | 62 | 17
  Adverse Event- Severe | 8 | 2
  Serious Adverse Event | 13 | 2
  Adverse Event leading to study medication discontinuation | 8 | 2

2. Secondary Outcome: Free Iscalimab Concentration in Plasma
Description: Free iscalimab concentration in plasma during the treatment (Ctrough) and follow-up (up to end of study) periods. Blood sample was collected at the specified timepoints to assess the concentration of free iscalimab. The baseline assessment of this extension study (Day 1) was identical to the last timepoint (FUP3/Week 60) of the core study (CCFZ533B2201).
Time Frame: Predose at Day 1, 113, 225, 337 and 421
Population: The pharmacokinetic set (PKS) included all participants who received at least one dose of iscalimab treatment and had quantifiable PK measurements of iscalimab. Number analysed refers to the number of participants with a quantifiable PK measurement at the specified time point
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram / mililiter
Arm/Group | Arm 1: Iscalimab 600 mg | Arm 2 - Iscalimab 300 mg
Number analyzed (Participants) | 149 | 52
microgram / mililiter
  Day 1 | 3.56 (372.2) | 451.8 (0.751)
  Day 113: number analyzed (Participants) | 137 | 50
  Day 113 | 125 (62.7) | 56.9 (54.0)
  Day 225: number analyzed (Participants) | 137 | 47
  Day 225 | 126 (104.7) | 50.3 (57.0)
  Day 337: number analyzed (Participants) | 107 | 37
  Day 337 | 138 (69.3) | 62.6 (63.3)
  Day 421: number analyzed (Participants) | 122 | 43
  Day 421 | 4.47 (533.7) | 350.4 (0.336)

3. Secondary Outcome: Incidence of Anti-iscalimab Antibodies in Plasma
Description: Number of participants with anti-iscalimab antibodies (ADA) in plasma at any time during the study. The baseline assessment of this extension study (Day 1) was identical to the last timepoint (FUP3/Week 60) of the core study (CCFZ533B2201).
Time Frame: 60 weeks
Population: The immunogenicity Set (IMS) included all subjects who received at least one dose of iscalimab treatment and had quantifiable immunogenicity measurements of iscalimab.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Iscalimab 600 mg | Arm 2 - Iscalimab 300 mg
Number analyzed (Participants) | 152 | 54
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: From start of extension study up to 14 weeks after last study-drug administration or end of study (whichever occurred earlier), assessed up to approximately 60 weeks
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up. The safety analysis were done on the safety population, which included all randomized subjects who received at least one dose of study medication. Patients were analyzed according to the actual treatment received.
Arm/Group | Arm 1: Iscalimab 600 mg | Arm 2 - Iscalimab 300 mg
All-Cause Mortality (participants affected / at risk) | 0/152 | 0/54
Serious Adverse Events (participants affected / at risk) | 13/152 | 2/54
Other Adverse Events (participants affected / at risk) | 102/152 | 38/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Iscalimab 600 mg (N=152) | Arm 2 - Iscalimab 300 mg (N=54)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Anal prolapse (Gastrointestinal disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Food allergy (Immune system disorders) | 1 | 0
Bartholinitis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Iscalimab 600 mg (N=152) | Arm 2 - Iscalimab 300 mg (N=54)
Neutropenia (Blood and lymphatic system disorders) | 10 | 2
Diarrhoea (Gastrointestinal disorders) | 13 | 4
Pyrexia (General disorders) | 8 | 2
COVID-19 (Infections and infestations) | 39 | 16
Influenza (Infections and infestations) | 7 | 7
Nasopharyngitis (Infections and infestations) | 22 | 9
Oral herpes (Infections and infestations) | 7 | 3
Sinusitis (Infections and infestations) | 7 | 3
Upper respiratory tract infection (Infections and infestations) | 19 | 5
Urinary tract infection (Infections and infestations) | 16 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 3
Headache (Nervous system disorders) | 9 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT04541589/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT04541589/SAP_001.pdf